CLINICAL TRIAL: NCT01754753
Title: Evaluation of the Effectiveness and Cost Effectiveness of an Intervention to Promote Mental Wellbeing in Community Living Older People.
Brief Title: Putting Life in Years (PLINY): Telephone Friendship Groups Research Study
Acronym: PLINY
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Due to lack of volunteer facilitators to deliver the intervention
Sponsor: University of Sheffield (Other)
Collaborators: University of Southampton (Other); Northumbria University (Other); Bangor University (Other); Age UK (Other); Community Network (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 09-3004-01; 28645428 (Registry Identifier: ISRCTN)
Record Dates: First submitted 2012-12-12; First posted 2012-12-21 (Estimated); Results first posted 2021-02-01 (Actual); Last update posted 2021-02-23 (Actual); Status verified 2016-05

CONDITIONS: Self Efficacy; Loneliness
Keywords: Mental well-being; Befriending
MeSH Terms: conditions — Psychological Well-Being

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Telephone friendship groups (Active Comparator): Participants allocated to telephone friendship groups will take part in 12 weekly group telephone discussions. The participant will be called, by a trained Age UK Sheffield volunteer, in their own home. The group discussions will take place for about an hour each week and involve between 6-8 participants. Participants will be introduced to weekly group calls by the volunteer who will call each participant individually for around 20 minutes each week for up to six weeks before the group is established.
  The group may have a particular focus or talk about different topics each week. The individual participants are joined together through a teleconferencing system (provided by Community Network).
  Interventions: Other: Telephone Friendship groups
- Usual health and social care (No Intervention): Participants allocated to the control arm will not receive any research intervention. However, they will participate in the research by completing questionnaires about their health and wellbeing.

INTERVENTIONS:
Other: Telephone Friendship groups
  Arms: Telephone friendship groups

SUMMARY:
The National Institute for Health Research commissioned this research with the following research question: "What is the relative effectiveness and cost effectiveness of home based support programmes in improving the mental wellbeing of older people living in their own homes?"

The project will evaluate whether telephone friendship groups, delivered by the voluntary sector over the telephone, can improve the mental wellbeing of older people aged 75 or over.

The research will also:

1. Identify the psychosocial and environmental factors, as well as implementation issues that may mediate or modify the effectiveness of the intervention using qualitative methods. This will include examining: 1.1. Assess voluntary sector readiness to take forward new forms of services; 1.2. The best modes of delivery of telephone support/friendship; 1.3. Assess how volunteers (facilitators) can be supported and retained; and, 1.4. The extent to which fidelity of the intervention is maintained within and across the participating organisations.
2. Determine if there is any lasting impact upon mental wellbeing by repeat measurement with all participants 12 months following baseline measurement
3. Examine whether there is any significant improvement on the physical dimension of the SF-36 at 6 months and 12 months, following baseline measure, for the intervention arm compared with usual care.
4. Measure the extent of use of health and social care, and community facilities by participants over time to determine whether the intervention is cost effective compared with usual care.

DETAILED DESCRIPTION:
Background and study aims:

People are living longer and many experience a good old age. Unfortunately longer life is not always accompanied by health and wellbeing. Older people can become lonely, isolated and unhappy as a result of a whole number of factors such as diminished physical abilities and bereavement.

Our research programme is examining how people aged 75 years and over can be helped to retain wellbeing and not feel unhappy due to feelings of loneliness and isolation. It is examining the possible benefits of group friendship over the telephone. Telephone befriending services are usually provided through the voluntary sector and are available in a number of locations. Befriending can take place on a one-to-one basis or through small groups of people linked together by telephone (teleconferencing). A small amount of research has already been conducted into telephone befriending. It appears to provide benefit but intevestigators need evidence from more people who have experienced befriending by telephone to be able to make clear statements about whether it should be recommended.

What does the study involve? To ensure that the research is thorough investigators want to recruit and involve 248 older people aged 75 years and over who live in Sheffield. It will take us over a year to recruit the number of older people investigators need as the befriending services can only accommodate a certain number of people at any one time.

The main method of inviting people to participate in the research is through letters of invitation from primary care. However investigators are also using other ways to get the information to those who might be interested such as giving talks at community venues and asking health and social care professionals to identify people who they think might benefit.

Everyone who has volunteered and is eligible to take part is randomly allocated to one of two groups. Not everyone will receive the research intervention (telephone friendship). Everyone is then asked questions about their wellbeing and health when they first meet a researcher and once again six months later. The investigators will compare the results from responses collected at the start of the study with the results collected six months later. The investigators will look to see whether those involved in telephone friendship groups feel happier about their lives compared with the group who were allocated to help in the research by answering questions only. To find out whether there might be any lasting benefit investigators will then ask all participants the same questions for a final time about 12 months after the start.

Those people allocated to receive telephone friendship will firstly receive up to six one-to-one calls from a trained and Criminal Records Bureau (CRB) checked Age UK Sheffield volunteer. The volunteer will talk to the participant for approximate 20 minutes and introduce them to the idea of group discussions over the telephone. They will then be invited to join a telephone friendship group with around six to seven other people. The friendship group then talk once a week for about one hour for 12 weeks with the group being assisted by an Age UK Sheffield volunteer.

As telephone friendship/ befriending services are relatively new, the investigators will look to see how they are being delivered and how people experience the service by talking with a small number of people have participated in the telephone friendship group. The investigators will also interview the Age UK Sheffield volunteers to find out if the telephone friendship service delivered to older people was as the investigators intended.

Older people are also helping us with the management of the study and continue to give their views on the progress of the project and any information that is being prepared. This is helping the researchers to ensure that what investigators ask people to do and any written material produced can be easily understood and meets the needs and expectations of those who are invited to take part.

Where is the study run from? The study is being organized by the University of Sheffield in partnership with Age UK and Community Network.

When is study starting and how long is it expected to run for? The study started on 1 October 2012 with invitations to join the study starting in June 2012 and continuing until May 2013. The study will run until December 2014 to enable us to follow-up participants, analyze the results and write a report of our findings.

Who is funding the study? National Institute for Health Research (NIHR), Public Health Research programme.

ELIGIBILITY:
Inclusion Criteria:

* Aged 75 years or over
* Good cognitive function, defined as Six Cognitive Impairment Test Brooke P, Bullock R, 1999) score of 7 or under;
* Living independently (including those who are co-resident with others) or in sheltered/ extra care housing;
* Able to understand and converse in English.

Exclusion Criteria:

* Aged 74 years or younger
* 6CIT score of 8 or more
* In residential/ nursing care homes
* Unable to understand and converse in English
* Unable to converse on the telephone with assertive technology 6. Already receiving a telephone intervention

Min Age: 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 157 (Actual)
Dates: Start 2012-06; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gail A Mountain, Principal Investigator — University of Sheffield
Locations (1):
- The University of Sheffield, Sheffield, United Kingdom

REFERENCES:
- See also: Click here for more information about this study — http://www.shef.ac.uk/scharr/sections/dts/ctru/pliny

RESULTS

PARTICIPANT FLOW:
Groups:
- Telephone Friendship Groups: Participants allocated to telephone friendship groups will take part in 12 weekly group telephone discussions. The participant will be called, by a trained Age UK Sheffield volunteer, in their own home. The group discussions will take place for about an hour each week and involve between 6-8 participants. Participants will be introduced to weekly group calls by the volunteer who will call each participant individually for around 20 minutes each week for up to six weeks before the group is established.
  The group may have a particular focus or talk about different topics each week. The individual participants are joined together through a teleconferencing system (provided by Community Network).
  Telephone Friendship groups
Period: Overall Study
Arm/Group | Telephone Friendship Groups | Usual Health and Social Care
Started | 78 | 79
Completed | 26 | 30
Not Completed | 52 | 49
Not completed — Study close | 43 | 44
Not completed — Lost to Follow-up | 9 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Telephone Friendship Groups | Usual Health and Social Care | Total
Number analyzed (Participants) | 78 | 79 | 157
Age, Continuous [Mean (Standard Deviation); unit: years] | 81.4 (4.9) | 80.3 (4.3) | 80.8 (4.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 54 | 51 | 105
  Male | 24 | 28 | 52
Race/Ethnicity, Customized [Number; unit: participants]
  English/Welsh/Scottish/Northern Irish/British | 74 | 74 | 148
  Any other white background | 1 | 4 | 5
  Carribbean | 1 | 0 | 1
  Indian | 0 | 1 | 1
  Irish | 1 | 0 | 1
  Prefer not to say | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: SF-36 Mental Health Dimension
Description: The Short Form 36 Health Survey Questionnaire (SF-36) is a 36 item scale, which measures eight domains of health status: physical functioning (10 items); physical role limitations (four items); bodily pain (two items); general health perceptions (five items); energy/vitality (four items); social functioning (two items); emotional role limitations (three items) and mental health (five items). A scoring algorithm is used to convert the raw scores into the eight dimensions listed above. The scores are transformed to range from zero where the respondent has the worst possible health to 100 where the respondent is in the best possible health.
Time Frame: SF36 at 6 months
Population: Intention to treat
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Telephone Friendship Groups | Usual Health and Social Care
Number analyzed (Participants) | 26 | 30
units on a scale | 77.5 (18.4) | 70.7 (21.2)

2. Secondary Outcome: Other Dimensions of the SF-36 (and Specifically Physical Health)
Description: as for outcome 1
Time Frame: SF36 other dimensions at 6 months
Population: Intention to treat
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Telephone Friendship Groups | Usual Health and Social Care
Number analyzed (Participants) | 26 | 30
units on a scale | 60.3 (29.9) | 56 (29.9)

3. Secondary Outcome: EQ-5D for Health Economic Analysis
Description: EuroQol-5D-3L (EQ-5D-3L) is an instrument which evaluates the generic quality of life developed in Europe and widely used. The EQ-5D descriptive system is a preference-based HRQL measure with one question for each of the five dimensions that include mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. This ranges from 1 (good health) to - 0.56.
Time Frame: EQ-5D at 6 months
Population: Intention to treat
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Telephone Friendship Groups | Usual Health and Social Care
Number analyzed (Participants) | 26 | 29
units on a scale | 0.73 (0.35) | 0.71 (0.27)

4. Secondary Outcome: General Perceived Self Efficacy (GSE) Scale
Description: The General Perceived Self Efficacy (GSE) Scale is a 10-item questionnaire assessing a person's coping resources. Responses are made on a 4-point scale. Summing up the responses to all 10 items yields the final composite score with a range from 10 to 40. Higher scores indicate higher perceived general self-efficacy, lower scores indicate lower perceived general self-efficacy
Time Frame: GSE at 6 months
Population: Intention to treat
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Telephone Friendship Groups | Usual Health and Social Care
Number analyzed (Participants) | 26 | 30
units on a scale | 32.9 (4.7) | 32.1 (3.8)

5. Secondary Outcome: Patient Health Questionnaire (PHQ-9)
Description: The Patient Health Questionnaire (PHQ)-9 is the major depressive disorder (MDD) module of the full PHQ. It scores each of the 9 DSM criteria of MDD as "0" (not at all) to "3" (nearly every day), providing a 0-27 severity score. Higher scores indicate better outcome.
Time Frame: PHQ-9 at 6 months
Population: Intention to treat
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Telephone Friendship Groups | Usual Health and Social Care
Number analyzed (Participants) | 26 | 30
units on a scale | 3.1 (4) | 3.6 (4.6)

6. Secondary Outcome: De Jong Loneliness Scale
Description: The de Jong Gierveld Loneliness Scale score is a measuring instrument for loneliness. The total scale score is the sum of the item scores, ranging from 0 (not lonely) to 11 (extremely lonely).
Time Frame: De Jong at 6 months
Population: Intention to treat
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Telephone Friendship Groups | Usual Health and Social Care
Number analyzed (Participants) | 26 | 30
units on a scale | 3.5 (3.4) | 3.3 (2.9)

7. Secondary Outcome: ONS Wellbeing Question
Description: The Office for National Statistics Wellbeing Question is a standard question used by Office for National Statistics to examine subjective wellbeing of the general population in the UK, with questions grouped in three domains - (evaluative, experience and eudemonic). It is scored on a 0 to 10 scale with a higher score indicating better well-being.
Time Frame: ONS wellbeing at 6 months
Population: Intention to treat
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Telephone Friendship Groups | Usual Health and Social Care
Number analyzed (Participants) | 26 | 30
units on a scale | 8 (1.5) | 7.6 (1.8)

ADVERSE EVENTS:
Time Frame: 6 months
Description: Six month follow-up data was collected by a research assistant via telephone. Follow up data involved the completion of the a checklist that elicited whether any serious events had occurred since baseline (life-threatening event, event requiring inpatient hospitalization or prolonging existing hospitalization, event resulting in persistent or significant disability/incapacity).
Arm/Group | Telephone Friendship Groups | Usual Health and Social Care
All-Cause Mortality (participants affected / at risk) | 0/78 | 0/79
Serious Adverse Events (participants affected / at risk) | 0/78 | 0/79
Other Adverse Events (participants affected / at risk) | 0/78 | 0/79

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No